CLINICAL TRIAL: NCT05703802
Title: Establishment of an Enzyme-linked Immunosorbent Assay for the Recognition of Procalcitonin Variants and Characterization of Procalcitonin Variants in Patients With Hyperprocalcitonemia.
Brief Title: Establishment of an ELISA for the Recognition of Procalcitonin Variants in Patients With Hyperprocalcitonemia.
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Sebastian Kintrup, Principal Investigator, University Hospital Muenster
Other Study IDs: 10-AnIt-19
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Sepsis; Pre-Eclampsia; Granulomatosis With Polyangiitis; Microscopic Polyangiitis; Adiposity; SIRS; Procalcitonin
MeSH Terms: conditions — Sepsis; Pre-Eclampsia; Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Sepsis: Withdrawal of 3 blood collection tubes for ELISA-measurements at a single time during hyperprocalcitoninemia.
  Interventions: Diagnostic Test: Procalcitonin-variants ELISA-Assay
- SIRS: Withdrawal of 3 blood collection tubes for ELISA-measurements at a single time during hyperprocalcitoninemia.
  Interventions: Diagnostic Test: Procalcitonin-variants ELISA-Assay
- Adiposity: Withdrawal of 3 blood collection tubes for ELISA-measurements at a single time during hyperprocalcitoninemia.
  Interventions: Diagnostic Test: Procalcitonin-variants ELISA-Assay
- Granulomatosis with polyangiitis / microscopic polyangiitis: Withdrawal of 3 blood collection tubes for ELISA-measurements at a single time during hyperprocalcitoninemia.
  Interventions: Diagnostic Test: Procalcitonin-variants ELISA-Assay
- Pre-eclampsia: Withdrawal of 3 blood collection tubes for ELISA-measurements at a single time during hyperprocalcitoninemia.
  Interventions: Diagnostic Test: Procalcitonin-variants ELISA-Assay
- Healthy controls: Withdrawal of 3 blood collection tubes for ELISA-measurements at a single time during hyperprocalcitoninemia.
  Interventions: Diagnostic Test: Procalcitonin-variants ELISA-Assay

INTERVENTIONS:
Diagnostic Test: Procalcitonin-variants ELISA-Assay — Observational study measuring procalcitonin-variants in different patient collectives by obtaining 3 blood collection tubes per patient.

SUMMARY:
Procalcitonin is a protein consisting of 116 amino-acids which can rapidly rise under inflammatory conditions and sepsis. More than 20 years ago it has been shown that dipeptidylpeptidase-4 (DPP-4) cleaves procalcitonin from the n-terminus, resulting in a truncated procalcitonin-variant which consists of 114 aminoacids. Within their workgroup the investigators found that the truncated procalcitonin-variant had deleterious effects on vascular integrity during sepsis in mice. However, it is unknown if this applies also in humans. By using an ELISA-assay the investigators want to examine the ratio between native and truncated human procalcitonin during diseases accompanied with hyperprocalcitoninemia and correlate the results with clinical data.

DETAILED DESCRIPTION:
Procalcitonin is a protein consisting of 116 amino-acids which can rapidly rise under inflammatory conditions and sepsis. More than 20 years ago it has been shown that dipeptidylpeptidase-4 (DPP-4) cleaves procalcitonin from the n-terminus, resulting in a truncated procalcitonin-variant which consists of 114 aminoacids.

Within their workgroup the investigators found that the truncated procalcitonin-variant had deleterious effects on vascular integrity during sepsis in mice: They observed that binding of truncated procalcitonin to the CRLR/RAMP1-receptor on vascular endothelium lead to phosphorylation and destruction of VE-cadherin, an essential part of adherens junctions. Consequently, paracellular leakage of proteins and fluid from blood vessels developed.

It is unknown if these effects also apply to humans. By using an ELISA-assay the investigators want to examine the ratio between native and truncated human procalcitonin during diseases accompanied with hyperprocalcitoninemia and correlate the results with clinical data. Futhermore, they want to examine if the procalcitonin-variants have influence on cytokine levels and surface antigens on immune cells by performing multiplex immunoassays and FACS-analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Patients with diagnosis...
* Sepsis or,
* SIRS after cardiothoracic surgery or,
* adipositas or,
* granulomatosis with polyangiitis/microscopic polyangiitis or,
* pre-eclampsia
* healthy control subjects
* written informed consent

Exclusion Criteria:

* participation in an interventional study trial within the last 3 months
* relationship to study investigator

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients from the University Hospital Münster who suffer from different diseases which are accompanied by hyperprocalcitoninemia.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Ratio between native and truncated procalcitonin during different conditions of hyperprocalcitoninemia | Blood withdrawal takes approximately 5 minutes per patient
  Measurement performed by using ELISA-assay.

SECONDARY OUTCOMES:
DPP-4-activity | Blood withdrawal takes approximately 5 minutes per patient
  Measurement performed by using a commercial DPP4-ELISA-kit.
Proinflammatory cytokines | Blood withdrawal takes approximately 5 minutes per patient
  Measurement performed by using a commercial multiplex immunoassay kit.
Immun cell surface-antigens | Blood withdrawal takes approximately 5 minutes per patient
  Measurement performed by using fluorescence-acivated cell sorting (FACS).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Münster, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wrenger S, Kahne T, Bohuon C, Weglohner W, Ansorge S, Reinhold D. Amino-terminal truncation of procalcitonin, a marker for systemic bacterial infections, by dipeptidyl peptidase IV (DP IV). FEBS Lett. 2000 Jan 21;466(1):155-9. doi: 10.1016/s0014-5793(99)01779-2. PMID 10648832
- [Background] Brabenec L, Muller M, Hellenthal KEM, Karsten OS, Pryvalov H, Otto M, Holthenrich A, Matos ALL, Weiss R, Kintrup S, Hessler M, Dell'Aquila A, Thomas K, Nass J, Margraf A, Nottebaum AF, Rossaint J, Zarbock A, Vestweber D, Gerke V, Wagner NM. Targeting Procalcitonin Protects Vascular Barrier Integrity. Am J Respir Crit Care Med. 2022 Aug 15;206(4):488-500. doi: 10.1164/rccm.202201-0054OC. PMID 35699655
- [Result] Weglohner W, Struck J, Fischer-Schulz C, Morgenthaler NG, Otto A, Bohuon C, Bergmann A. Isolation and characterization of serum procalcitonin from patients with sepsis. Peptides. 2001 Dec;22(12):2099-103. doi: 10.1016/s0196-9781(01)00541-1. PMID 11786196
- [Derived] Kintrup S, Brabenec L, Zurek-Leffers FM, Hellenthal KEM, Cyran L, Meybohm P, Gerke V, Wagner NM. Detection and Evaluation of Procalcitonin Variants As Diagnostic Tools in Systemic Inflammation. Anesth Analg. 2025 May 1;140(5):1073-1082. doi: 10.1213/ANE.0000000000007170. PMID 39636188